CLINICAL TRIAL: NCT02153944
Title: Cognitive vs. Emotional Psycho-Pharmacological Manipulations of Fear vs. Anxiety
Brief Title: Cognitive vs. Emotional Psychopharmacological Manipulations of Fear vs. Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 140114; 14-M-0114
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Results first posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2021-10

CONDITIONS: Anxiety Disorder
Keywords: Startle; Induced-Threat; Memory; Stimulant; Cognitive Interference
MeSH Terms: conditions — Anxiety Disorders | interventions — Propranolol; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Behavioral: Drug challenge with methylphenidate (Experimental): Participant received methylphenidate 20 mg orally during study visit
  Interventions: Drug: Methylphenidate
- Behavioral: Drug challenge with placebo (Placebo Comparator): Participant received placebo orally during study visit
  Interventions: Drug: Placebo
- Behavioral: Drug challenge with propranolol (Experimental): Participants received propranolol 40mg orally during study visit
  Interventions: Drug: Propranolol
- fMRI: Drug challenge with methylphenidate (Experimental): Participant received methylphenidate 20 mg orally during study visit
  Interventions: Drug: Methylphenidate
- fMRI: Drug challenge with placebo (Placebo Comparator): Participant received placebo orally during study visit
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Propranolol 40 mg was given orally during study visit
  Arms: Behavioral: Drug challenge with propranolol
Drug: Methylphenidate — Methylphenidate 20mg was given orally during study visit
  Arms: Behavioral: Drug challenge with methylphenidate; fMRI: Drug challenge with methylphenidate
Drug: Placebo — Placebo was given orally during study visit
  Arms: Behavioral: Drug challenge with placebo; fMRI: Drug challenge with placebo

SUMMARY:
Objective:

The overall aim of this protocol is to examine the effect of pharmacological manipulations of affective and cognitive processes on anxiety and task performance. Ultimately, the goal is 1) to provide insight into the relative influence of cognitive and affective states on anxiety, 2) generate theoretical models that can be applied to a better understanding of the interaction between cognition and emotion, 3) develop a better screening approach to candidate anxiolytics, and 4) help formulate novel therapeutic interventions for clinical anxiety.

Excessive or inappropriately sustained anxiety and fear lead to the most common group of psychiatric disorders. A number of theoretical models have been proposed to understand the mechanisms engaged in these maladaptive behaviors. Most recent emphasis has focused on the synergistic contribution of cognitive and emotional processes. Our laboratory has been instrumental in delineating aspects of behavioral and neural processes that are associated with fear and anxiety, using psychophysiological and neuroimaging measures of fear and anxiety. Evidence shows that levels of anxiety modulate cognitive performance, such as working memory or perceptual discrimination, and that, conversely, cognitive engagement influences severity of experimentally induced anxiety. The exact contribution of emotional processes vs. cognitive processes to the experience of anxiety is not clear, similarly to the neural mechanisms underlying these interactions.

In this protocol, we propose to manipulate pharmacologically separately cognitive and emotional processes to dissociate their contribution to fear/anxiety, while using state-of-the-art measures of anxiety derived from translational work. Indeed, we already developed integrative experimental models of fear and anxiety via the manipulation of predictable and unpredictable shock, respectively. We already employed successfully these models to measure anxiolytic and anxiogenic effects of various compounds such as alprazolam, citalopram, hydrocortisone, and oxytocin in healthy participants.

We propose in a first step (step-1) to start with a simple proof-of-concept study, using two pharmacological compounds in a double-blind randomized parallel design, each preferentially acting respectively on the cognitive (methylphenidate) or affective (propranolol) domain, and using a single cognitive process (working memory). In a second step (step-2), we propose to extend this work to the fMRI to examine the cognitive correlates of the effects seen in the step-1 behavioral study, specifically with methylphenidate. Whereas the comparison among three drugs is planned for the electrophysiology study, we plan to study only the drug that improves cognition in the fMRI. The reason we will focus on methylphenidate in step 2 is that our overall goal is to study the effect of improving cognitive functions on anxiety using neuroimaging. To reach this goal, we plan to use different approaches to boost cognitive functions in the coming years, including psychopharmacology, direct current stimulation, mindfulness. Methylphenidate is our first psychopharmacological study towards this objective. Future work will also expand to other compounds and cognitive processes, as well as vary the strategy to induce anxiety. Presently, anxiety will be induced using the threat of shock, while participants perform the task. We will examine in step-1 whether 1) the reduction of induced-anxiety with propranolol improves cognitive performance, and 2) the facilitation of cognitive performance with methylphenidate reduces induced-anxiety. In step-2, we will identify the neural mechanisms underlying the effects of methylphenidate, the drug having beneficial effects on cognitive function.

Study population:

Medically and psychiatrically healthy adult males and females, aged 18 to 50 years.

Design:

The study is a double-blind design. For step-1, three groups of healthy participants will come for one experimental session. During this session, they will be asked to perform a working memory task under the threat of shock, i.e., while anticipating unpleasant electric shocks. Each group will receive one drug challenge, either placebo, propranolol (40 g) or methylphenidate (20 mg). For step-2, the study tasks will be conducted in a 3T fMRI scanner. In this step, only methylphenidate and placebo will be compared. Two groups will come for one experimental session, one will receive placebo and the other one will receive methylphenidate (20 mg). In a follow-up study for the step-2 fMRI the two groups will come for one experimental fMRI session one will receive methylphenidate (60 mg).

Outcome measures:

In step-1, the primary outcome measures are the startle reflex and performance on the working memory task. In step-2, the primary outcome measures are the startle reflex and the cerebral fMRI blood-oxygen-level ...

DETAILED DESCRIPTION:
Objective:

The overall aim of this protocol is to examine the effect of pharmacological manipulations of affective and cognitive processes on anxiety and task performance. Ultimately, the goal is 1) to provide insight into the relative influence of cognitive and affective states on anxiety, 2) generate theoretical models that can be applied to a better understanding of the interaction between cognition and emotion, 3) develop a better screening approach to candidate anxiolytics, and 4) help formulate novel therapeutic interventions for clinical anxiety.

Excessive or inappropriately sustained anxiety and fear lead to the most common group of psychiatric disorders. A number of theoretical models have been proposed to understand the mechanisms engaged in these maladaptive behaviors. Most recent emphasis has focused on the synergistic contribution of cognitive and emotional processes. Our laboratory has been instrumental in delineating aspects of behavioral and neural processes that are associated with fear and anxiety, using psychophysiological and neuroimaging measures of fear and anxiety. Evidence shows that levels of anxiety modulate cognitive performance, such as working memory or perceptual discrimination, and that, conversely, cognitive engagement influences severity of experimentally induced anxiety. The exact contribution of emotional processes vs. cognitive processes to the experience of anxiety is not clear, similarly to the neural mechanisms underlying these interactions.

In this protocol, we propose to manipulate pharmacologically separately cognitive and emotional processes to dissociate their contribution to fear/anxiety, while using state-of-the-art measures of anxiety derived from translational work. Indeed, we already developed integrative experimental models of fear and anxiety via the manipulation of predictable and unpredictable shock, respectively. We already employed successfully these models to measure anxiolytic and anxiogenic effects of various compounds such as alprazolam, citalopram, hydrocortisone, and oxytocin in healthy participants.

We propose in a first step (step-1) to start with a simple proof-of-concept study, using two pharmacological compounds in a double-blind randomized parallel design, each preferentially acting respectively on the cognitive (methylphenidate) or affective (propranolol) domain, and using a single cognitive process (working memory). In a second step (step-2), we propose to extend this work to the fMRI to examine the cognitive correlates of the effects seen in the step-1 behavioral study, specifically with methylphenidate. Whereas the comparison among three drugs is planned for the electrophysiology study, we plan to study only the drug that improves cognition in the fMRI. The reason we will focus on methylphenidate in step 2 is that our overall goal is to study the effect of improving cognitive functions on anxiety using neuroimaging. To reach this goal, we plan to use different approaches to boost cognitive functions in the coming years, including psychopharmacology, direct current stimulation, mindfulness. Methylphenidate is our first psychopharmacological study towards this objective. Future work will also expand to other compounds and cognitive processes, as well as vary the strategy to induce anxiety. Presently, anxiety will be induced using the threat of shock, while participants perform the task. We will examine in step-1 whether 1) the reduction of induced-anxiety with propranolol improves cognitive performance, and 2) the facilitation of cognitive performance with methylphenidate reduces induced-anxiety. In step-2, we will identify the neural mechanisms underlying the effects of methylphenidate, the drug having beneficial effects on cognitive function.

Study population:

Medically and psychiatrically healthy adult males and females, aged 18 to 50 years.

Design:

The study is a double-blind design. For step-1, three groups of healthy participants will come for one experimental session. During this session, they will be asked to perform a working memory task under the threat of shock, i.e., while anticipating unpleasant electric shocks. Each group will receive one drug challenge, either placebo, propranolol (40 g) or methylphenidate (20 mg). For step-2, the study tasks will be conducted in a 3T fMRI scanner. In this step, only methylphenidate and placebo will be compared. Two groups will come for one experimental session, one will receive placebo and the other one will receive methylphenidate (20 mg). In a follow-up study for the step-2 fMRI the two groups will come for one experimental fMRI session one will receive methylphenidate (60 mg).

Outcome measures:

In step-1, the primary outcome measures are the startle reflex and performance on the working memory task. In step-2, the primary outcome measures are the startle reflex and the cerebral fMRI blood-oxygen-level dependent (BOLD) responses. For both step-1 and step-2, secondary measures include skin conductance, heart rate, and subjective measures of anxiety.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ages 18-50
* Males and females
* Subjects give their own consent

EXCLUSION CRITERIA:

* Clinically significant prior exposure to medications, that based on the investigator s judgment, may impact the study, such as Ritalin (MPH).
* Any significant medical or neurological problems (e.g. cardiovascular illness, respiratory illness, neurologic illness, seizure, etc.)
* Raynaud syndrome
* IQ < 80
* Sinus bradycardia (P<45), or tachycardia (P>90)
* Significant ECG abnormality (i.e., greater than first-degree block etc.) as determined by investigators judgement
* High or low blood pressure (SBP>140 or SBP<90; SDP<50 or SDP>90)
* A first-degree family history of mania, schizophrenia, or other psychoses based on verbal reports
* Significant past psychopathology (e.g., hospitalization for psychiatric disorders, recurrent depression, suicide attempt, psychoses)
* Current psychiatric disorders according to Diagnostic and Statistical Manual (DSM)-V
* Current alcohol or substance use disorder
* Current use of psychotropic medication
* Impaired hearing (clinic study only)
* Pregnancy or positive pregnancy test
* Neurological syndrome of the wrist (e.g., carpal tunnel syndrome) for shocks to be delivered on affected arm.
* Breastfeeding
* Significant lab abnormalities (i.e., complete blood count (CBC) with differential, acute care and mineral panel, hepatic panel, TSH)
* Positive urine toxicology screen
* You have been in another study with an experimental medication within the previous month
* For physiological/clinic participants: small startle reactivity (a change in EMG activity that is less than 3 times the baseline EMG activity)
* Current daily use of anti-acid -medication or within 5 half-lives of study visit if taken on pro re nata (PRN) basis
* Employee of National Institute of Mental Health (NIMH) or an immediate family member who is a NIMH employee.
* For functional magnetic resonance imaging (fMRI) participants: Any medical condition that increases risk for fMRI:

  * Any metal implants (clips, screws, plates, pins, etc.) that are not safe for MRI or metal fragments cause by injuries or metal working. Metal implants that are deemed MRI safe are allowable (i.e. certain screws).
  * Any sort of medical implants that are not safe for the MRI (aneurysm clips, pacemaker, insulin pump, Hickman line, etc.). Medical implants that are MRI safe (Nexplanon implant, certain intrauterine device (IUDs), etc.) are allowable.
  * Permanent eye liner and tattoos above the neck
  * Patients who have difficulty lying flat on their back for up to 90 min in the scanner
  * Participants who are uncomfortable in small closed spaces (have claustrophobia) and would feel uncomfortable in the MRI machine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monique Ernst, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Gaillard C, Lago TR, Gorka AX, Balderston NL, Fuchs BA, Reynolds RC, Grillon C, Ernst M. Methylphenidate modulates interactions of anxiety with cognition. Transl Psychiatry. 2021 Oct 21;11(1):544. doi: 10.1038/s41398-021-01621-2. PMID 34675189
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-M-0114.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 participants who signed consent did not meet the inclusion criteria so were excluded from study
Pre-assignment Details: Total of 142 unique subjects were consented to this protocol. One subject from the Behavioral study also participated in the fMRI: Drug Challenge With Placebo.
Groups:
- fMRI: Drug Challenge With Methylphenidate: Participant received methylphenidate 20 mg orally during a single day six hour study visit
- fMRI: Drug Challenge With Placebo: Participant received placebo orally during a single day six hour study visit
Period: Behavioral Sub-study
Arm/Group | Behavioral: Drug Challenge With Methylphenidate | Behavioral: Drug Challenge With Placebo | Behavioral: Drug Challenge With Propranolol | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Started | 20 | 20 | 20 | 0 | 0
Completed | 20 | 20 | 20 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: fMRI Sub-study
Arm/Group | Behavioral: Drug Challenge With Methylphenidate | Behavioral: Drug Challenge With Placebo | Behavioral: Drug Challenge With Propranolol | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Started | 0 | 0 | 0 | 34 | 35 (Include one subject from Behavioral: Drug challenge with propranolol)
Completed | 0 | 0 | 0 | 34 | 35
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject from the Behavioral study also participated in the fMRI: Drug Challenge With Placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral: Drug Challenge With Methylphenidate | Behavioral: Drug Challenge With Placebo | Behavioral: Drug Challenge With Propranolol | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo | Total
Number analyzed (Participants) | 20 | 20 | 20 | 34 | 34 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 34 | 34 | 128
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 18 | 18 | 66
  Male | 10 | 10 | 10 | 16 | 16 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 4 | 3 | 10 | 20
  Not Hispanic or Latino | 19 | 18 | 16 | 31 | 24 | 108
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 2 | 3 | 2 | 8 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 4 | 9 | 10 | 32
  White | 11 | 11 | 12 | 14 | 15 | 63
  More than one race | 3 | 0 | 0 | 2 | 1 | 6
  Unknown or Not Reported | 0 | 1 | 2 | 1 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of Startle Reflex During Safe Condition
Description: The magnitude of the startle reflex during working memory tasks (n-back) while undergoing alternating periods of safety and threat of shock. The n-back is a paradigm used to assess working memory function by presenting sequential stimuli individually. The participant holds each stimulus in short-term memory while new stimuli are presented. For each new item presented, the participant's task is to decide if it is the same as the stimulus presented one time before (1Back), two times before (2Back) or three times before (3Back) by responding "yes" if the stimulus currently presented matches the stimulus presented earlier. Participants responded with a button press. The startle reflex was elicited with a 102 decibel (dB) white noise (40-ms duration) delivered via headphone. The eyeblink component of the startle reflex was recorded binaurally with two silver chloride (AgCl) electrodes placed under one eye.
Time Frame: 20-120 milliseconds following the onset of the startle stimulus
Population: Analyses included subjects who completed the behavioral study arms.
Measure: Mean (Standard Error); unit: millivolts (mV)
Arm/Group | Behavioral: Drug Challenge With Methylphenidate | Behavioral: Drug Challenge With Placebo | Behavioral: Drug Challenge With Propranolol
Number analyzed (Participants) | 20 | 20 | 20
millivolts (mV)
  1Back | 42.2880893 (0.556162) | 42.39801 (0.471667) | 43.61243 (0.667329)
  2Back | 44.1886408 (0.441141) | 45.32989 (0.65412) | 44.96692 (0.37425)
  3Back | 45.7608354 (0.585204) | 46.63108 (0.663525) | 47.15858 (0.531088)

2. Primary Outcome: Magnitude of Startle Reflex During Threat Condition
Description: as for outcome 1
Time Frame: 20-120 milliseconds following the onset of the startle stimulus
Population: Analyses included subjects who completed the behavioral study arms.
Measure: Mean (Standard Error); unit: millivolts (mV)
Arm/Group | Behavioral: Drug Challenge With Methylphenidate | Behavioral: Drug Challenge With Placebo | Behavioral: Drug Challenge With Propranolol
Number analyzed (Participants) | 20 | 20 | 20
millivolts (mV)
  1Back | 51.6813833 (0.914442) | 51.79882 (0.789383) | 52.20783 (0.835526)
  2Back | 51.0953725 (0.714049) | 51.61492 (0.762457) | 50.13929 (0.719978)
  3Back | 52.1700802 (0.966944) | 51.40215 (0.875497) | 50.53474 (0.707909)

3. Primary Outcome: Proportion of Correct Responses in the Working Memory Task (N-back) - Safe Condition
Description: Stimuli were presented one at a time on a screen. Participants were instructed to remember (working memory) one, two, or three stimuli back (N-back) from the current stimulus on the screen while undergoing alternating periods of safety and threat of shock i.e. while anticipating unpleasant electric shocks or no shock (safe). The n-back is a paradigm used to assess working memory function by presenting sequential stimuli individually. The participant holds each stimulus in short-term memory while new stimuli are presented. For each new item presented, the participant's task is to decide if it is the same as the stimulus presented one time before (1Back), two times before (2Back) or three times before (3Back)" by responding "yes" if the stimulus currently presented matches the stimulus presented earlier. Performance on working memory task (n-back) accuracy was measured across condition (threat and safe) x Load (1Back, 2Back, 3Back) using repeated measures ANOVA.
Time Frame: Task started 90 minutes post drug admin up to max of 125 mins post drug admin (max total is 35 mins) during a 6-hour single day visit
Population: Analyses included subjects who completed the behavioral study arms.
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | Behavioral: Drug Challenge With Methylphenidate | Behavioral: Drug Challenge With Placebo | Behavioral: Drug Challenge With Propranolol
Number analyzed (Participants) | 20 | 20 | 20
Proportion of correct responses
  1Back | 0.96235 (0.006836) | 0.9285 (0.014375) | 0.94535 (0.012417)
  2Back | 0.92585 (0.019265) | 0.8734 (0.02145) | 0.9039 (0.018021)
  3Back | 0.82115 (0.024021) | 0.792 (0.022333) | 0.8528 (0.020582)

4. Primary Outcome: Proportion of Correct Responses in the Working Memory Task (N-back) - Threat Condition
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Analyses included subjects who completed the behavioral study arms.
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | Behavioral: Drug Challenge With Methylphenidate | Behavioral: Drug Challenge With Placebo | Behavioral: Drug Challenge With Propranolol
Number analyzed (Participants) | 20 | 20 | 20
Proportion of correct responses
  1Back | 0.9586 (0.012115) | 0.92755 (0.011995) | 0.94445 (0.014309)
  2Back | 0.88505 (0.020467) | 0.83255 (0.024274) | 0.88275 (0.018205)
  3Back | 0.8358 (0.025528) | 0.74575 (0.025876) | 0.8152 (0.018288)

5. Primary Outcome: Proportion of Correct Responses in the Working Memory Task (N-Back): Safe Condition - 1BACK - Run 1
Description: Stimuli were presented one at a time on a screen. Participants were instructed to remember (working memory) one or three stimuli back (N-back) from the current stimulus on the screen while undergoing alternating periods of safety and threat of shock i.e. while anticipating unpleasant electric shocks or no shock (safe).Two levels of difficulties were tested: 1- and 3-back. The n-back is a paradigm used to assess working memory function by presenting sequential stimuli individually. Participants indicated whether the letter currently displayed was the same as the letter presented 1 or 3 letters back. The task included 3 runs, 8 blocks per run (4 safe and 4 threat presented alternatively), 18 sequential letters per block. Each block represented a given level of difficulty, i.e., 1- and 3-back. Performance on working memory task (n-back) accuracy was measured across condition (threat and safe) x Load (1-back, 3-back) using repeated measures ANOVA.
Time Frame: 90 minutes post drug admin plus zero seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 32 | 33
Proportion of correct responses | 0.9565625 (0.0128155) | 0.919697 (0.0155851)

6. Primary Outcome: Proportion of Correct Responses in the Working Memory Task (N-back): Threat Condition - 1BACK - Run 1
Description: Stimuli were presented one at a time on a screen. Participants were instructed to remember (working memory) one or three stimuli back (N-back) from the current stimulus on the screen while undergoing alternating periods of safety and threat of shock i.e. while anticipating unpleasant electric shocks or no shock (safe). Two levels of difficulties were tested: 1- and 3-back. The n-back is a paradigm used to assess working memory function by presenting sequential stimuli individually. Participants indicated whether the letter currently displayed was the same as the letter presented 1 or 3 letters back. The task included 3 runs, 8 blocks per run (4 safe and 4 threat presented alternatively), 18 sequential letters per block. Each block represented a given level of difficulty, i.e., 1- and 3-back. Performance on working memory task (n-back) accuracy was measured across condition (threat and safe) x Load (1-back, 3-back) using repeated measures ANOVA.
Time Frame: 90 minutes plus 90 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 32 | 33
Proportion of correct responses | 0.9228125 (0.0116936) | 0.9378788 (0.0152737)

7. Primary Outcome: Proportion of Correct Responses in the Working Memory Task (N-back): Safe Condition - 1BACK - Run 2
Description: as for outcome 6
Time Frame: 90 minutes plus 180 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 31 | 32
Proportion of correct responses | 0.9529032 (0.0152273) | 0.953125 (0.0127193)

8. Primary Outcome: Proportion of Correct Responses in the Working Memory Task (N-back): Threat Condition - 1BACK - Run 2
Description: as for outcome 6
Time Frame: 90 minutes plus 260 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 31 | 32
Proportion of correct responses | 0.9435484 (0.0120353) | 0.9425 (0.0123703)

9. Primary Outcome: Proportion of Correct Responses in the Working Memory Task (N-back): Safe Condition - 3BACK - Run 1
Description: as for outcome 6
Time Frame: 90 minutes post drug admin plus 45 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 32 | 33
Proportion of correct responses | 0.725625 (0.0199543) | 0.739697 (0.0169418)

10. Primary Outcome: Proportion of Correct Responses in the Working Memory Task (N-back): Threat Condition - 3BACK - Run 1
Description: as for outcome 6
Time Frame: 90 minutes plus 135 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 32 | 33
Proportion of correct responses | 0.73 (0.0209454) | 0.7275758 (0.0173862)

11. Primary Outcome: Proportion of Correct Responses in the Working Memory Task (N-back): Safe Condition - 3BACK - Run 2
Description: as for outcome 6
Time Frame: 90 minutes plus 215 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 31 | 32
Proportion of correct responses | 0.7570968 (0.0203844) | 0.7428125 (0.0154713)

12. Primary Outcome: Proportion of Correct Responses in the Working Memory Task (N-back): Threat Condition - 3BACK - Run 2
Description: as for outcome 6
Time Frame: 90 minutes plus 305 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 31 | 32
Proportion of correct responses | 0.7816129 (0.0195767) | 0.7671875 (0.0212949)

13. Primary Outcome: Reaction Time to Stimuli: Safe Condition - 1BACK - Run 1
Description: Reaction time (RT) is the time it takes to respond to stimuli. Participants RTs were measured while undergoing alternating periods of safety and shock threat conditions i.e. while anticipating unpleasant electric shocks (threat) or no shock (safe) during the n-back paradigm task. The n-back is a paradigm used to assess working memory function by presenting sequential stimuli individually. Two levels of difficulties were tested: 1Back and 3Back (n-back). Participants were instructed to indicate whether the letter currently displayed was the same as the letter presented 1 or 3 letters back. The task was organized in 2 runs, 8 blocks per run (4 safe and 4 threat presented alternatively), 18 sequential letters per block. Each block (threat or safe) corresponded to 2 tasks, 1- and 3-back tasks. RT was analyzed using condition( threat, safe) x Load (1Back, 3Back) repeated-measures ANOVA.
Time Frame: 90 minutes post drug admin plus zero seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 32 | 33
milliseconds (ms) | 743.283125 (34.2610375) | 794.7833333 (25.5496031)

14. Primary Outcome: Reaction Time to Stimuli: Threat Condition - 1BACK - Run 1
Description: Reaction time (RT) is the time it takes to respond to stimuli. Participants RTs were measured while undergoing alternating periods of safety and shock threat conditions i.e. while anticipating unpleasant electric shocks (threat) or no shock (safe) during the n-back paradigm task. The n-back is a paradigm used to assess working memory function by presenting sequential stimuli individually. Two levels of difficulties were tested: 1Back and 3Back (n-back). Participants were instructed to indicate whether the letter currently displayed was the same as the letter presented 1 or 3 letters back. The task was organized in 2 runs, 8 blocks per run (4 safe and 4 threat presented alternatively), 18 sequential letters per block. Each block (threat or safe) corresponded to 2 tasks, 1- and 3-back tasks. RT was analyzed using condition (threat, safe) x Load (1Back, 3Back) repeated-measures ANOVA.
Time Frame: 90 minutes plus 90 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 32 | 33
milliseconds (ms) | 771.2671875 (31.1029031) | 779.1712121 (26.243248)

15. Primary Outcome: Reaction Time to Stimuli: Safe Condition - 1BACK - Run 2
Description: as for outcome 14
Time Frame: 90 minutes plus 180 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 31 | 32
milliseconds (ms) | 707.7925806 (32.3045364) | 741.5425 (24.3019917)

16. Primary Outcome: Reaction Time to Stimuli: Threat Condition - 1BACK - Run 2
Description: as for outcome 14
Time Frame: 90 minutes plus 260 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 31 | 32
milliseconds (ms) | 729.0251613 (35.0943102) | 735.5509375 (18.592916)

17. Primary Outcome: Reaction Time to Stimuli: Safe Condition - 3BACK - Run 1
Description: as for outcome 14
Time Frame: 90 minutes post drug admin plus 45 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 32 | 33
milliseconds (ms) | 976.1853125 (51.3801064) | 1007.74 (42.2557395)

18. Primary Outcome: Reaction Time to Stimuli: Threat Condition - 3BACK - Run 1
Description: as for outcome 14
Time Frame: 90 minutes plus 135 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 32 | 33
milliseconds (ms) | 971.676875 (54.0569586) | 995.619697 (40.0099943)

19. Primary Outcome: Reaction Time to Stimuli: Safe Condition - 3BACK - Run 2
Description: as for outcome 14
Time Frame: 90 minutes plus 215 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 31 | 32
milliseconds (ms) | 912.6574194 (57.9059418) | 915.005625 (43.335215)

20. Primary Outcome: Reaction Time to Stimuli: Threat Condition - 3BACK - Run 2
Description: as for outcome 14
Time Frame: 90 minutes plus 305 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 31 | 32
milliseconds (ms) | 925.3409677 (55.550186) | 929.6796875 (33.7722034)

21. Primary Outcome: Measure of BOLD Response in Brain Clusters - Safe Condition - 1BACK
Description: The blood-oxygen-level dependent (BOLD) responses were measured using an fMRI scanner. The cerebral fMRI BOLD uses magnetic fields to measure localized changes in brain blood flow and blood oxygenation in activated regions-of-interest (ROI). Participants BOLD responses were measured while undergoing alternating periods of safety and shock threat conditions i.e. while anticipating unpleasant electric shocks or no shock (safe) during the n-back task. The n-back is a paradigm used to assess working memory function by presenting sequential stimuli individually. Two levels of difficulties were tested: 1Back and 3Back (n-back). Participants were instructed to indicate whether the letter currently displayed was the same as the letter presented 1 or 3 letters back.
Time Frame: started 90 minutes post drug administration plus 90 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: arbitrary units (A.U)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 29 | 31
arbitrary units (A.U)
  Brain Cluster-001 - Posterior Cingulate Cortex (PCC) | -0.151002 (0.0183468) | -0.2039758 (0.0234864)
  Brain Cluster-002 - Right Prefrontal Cortex (PFC) | -0.0712797 (0.0141168) | -0.1167484 (0.0189171)
  Brain Cluster-003 - Left Prefrontal Cortex (PFC) | -0.1331336 (0.0171501) | -0.1876725 (0.0240544)
  Brain Cluster-004 - Anterior Cingulate Cortex (ACC) | -0.1140823 (0.0200346) | -0.151052 (0.0219622)
  Brain Cluster-009 - Right Putamen | -0.0501889 (0.0123786) | -0.0848515 (0.0152059)
  Brain Cluster-11 - Frontal Pole | -0.0928793 (0.0380362) | -0.0743447 (0.0233097)
  Brain Cluster-12 - Right Insula | -0.0349776 (0.0227349) | -0.0830865 (0.0141616)
  Brain Cluster-13 - Frontal Pole | -0.1301602 (0.0242121) | -0.1309601 (0.0221458)
  Brain Cluster-14 - Right Insula | -0.0431302 (0.0169232) | -0.0856204 (0.0135548)

22. Primary Outcome: Measure of BOLD Response in Brain Cluster - Threat Condition - 1BACK
Description: as for outcome 21
Time Frame: started 90 minutes post drug administration plus up to 360 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: arbitrary units (A.U)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 29 | 31
arbitrary units (A.U)
  Brain Cluster-001 - Posterior Cingulate Cortex (PCC) | -0.1725431 (0.0203001) | -0.1488312 (0.027668)
  Brain Cluster-002 - Right Prefrontal Cortex (PFC) | -0.0806112 (0.0151041) | -0.0609964 (0.0205423)
  Brain Cluster-003 - Left Prefrontal Cortex (PFC) | -0.1557721 (0.0183071) | -0.1297947 (0.027029)
  Brain Cluster-004 - Anterior Cingulate Cortex (ACC) | -0.1201138 (0.0213735) | -0.0940195 (0.0234725)
  Brain Cluster-009 - Right Putamen | -0.06733 (0.0112697) | -0.0435053 (0.016678)
  Brain Cluster-11 - Frontal Pole | -0.0929706 (0.0369173) | -0.0173495 (0.0212833)
  Brain Cluster-12 - Right Insula | -0.0543121 (0.0175828) | -0.0434811 (0.0156982)
  Brain Cluster-13 - Frontal Pole | -0.1420901 (0.030675) | -0.0822257 (0.0286209)
  Brain Cluster-14-Right Insula | -0.0580487 (0.0198727) | -0.0542862 (0.016025)

23. Primary Outcome: Measure of BOLD Response in Brain Clusters - Safe Condition - 3BACK
Description: The blood-oxygen-level dependent (BOLD) responses were measured using an fMRI scanner. The cerebral fMRI BOLD uses magnetic fields to measure localized changes in brain The blood-oxygen-level dependent (BOLD) responses were measured using an fMRI scanner. The cerebral fMRI BOLD uses magnetic fields to measure localized changes in brain blood flow and blood oxygenation in activated regions-of-interest (ROI). Participants BOLD responses were measured while undergoing alternating periods of safety and shock threat conditions i.e. while anticipating unpleasant electric shocks or no shock (safe) during the n-back task. The n-back is a paradigm used to assess working memory function by presenting sequential stimuli individually. Two levels of difficulties were tested: 1Back and 3Back (n-back). Participants were instructed to indicate whether the letter currently displayed was the same as the letter presented 1 or 3 letters back.
Time Frame: started 90 minutes post drug administration plus up to 270 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: arbitrary units (A.U)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 29 | 31
arbitrary units (A.U)
  Brain Cluster-001 - Posterior Cingulate Cortex (PCC) | -0.1255616 (0.0232653) | -0.1256943 (0.0246892)
  Brain Cluster-002 - Right Prefrontal Cortex (PFC) | -0.0557781 (0.0185596) | -0.0542905 (0.0175298)
  Brain Cluster-003 - Left Prefrontal Cortex (PFC) | -0.0797764 (0.0218839) | -0.0719455 (0.0222242)
  Brain Cluster-004 - Anterior Cingulate Cortex (ACC) | -0.1212111 (0.0251039) | -0.1206337 (0.0215921)
  Brain Cluster-009 - Right Putamen | -0.0716675 (0.0136668) | -0.0560306 (0.0157124)
  Brain Cluster-11 - Frontal Pole | -0.0695188 (0.0305467) | 0.001909 (0.0229718)
  Brain Cluster-12 - Right Insula | -0.0868275 (0.0233106) | -0.0971834 (0.0209667)
  Brain Cluster-13 - Frontal Pole | -0.2002039 (0.0345408) | -0.1695771 (0.029338)
  Brain Cluster-14 - Right Insula | -0.0783793 (0.0201576) | -0.0832567 (0.014176)

24. Primary Outcome: Measure of BOLD Response in Brain Cluster - Threat Condition - 3BACK
Description: as for outcome 21
Time Frame: started 90 minutes post drug administration plus up to 450 seconds within a 6-hour study visit
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: arbitrary units (A.U)
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 29 | 31
arbitrary units (A.U)
  Brain Cluster-001 - Posterior Cingulate Cortex (PCC) | -0.0884053 (0.0221989) | -0.1575204 (0.0247188)
  Brain Cluster-002 - Right Prefrontal Cortex (PFC) | -0.0248587 (0.0197718) | -0.0701165 (0.017604)
  Brain Cluster-003 - Left Prefrontal Cortex (PFC) | -0.0465762 (0.0236681) | -0.0900214 (0.0252627)
  Brain Cluster-004 - Anterior Cingulate Cortex (ACC) | -0.089146 (0.0262966) | -0.1278046 (0.0225001)
  Brain Cluster-009 - Right Putamen | -0.0470163 (0.0185279) | -0.0758935 (0.0144397)
  Brain Cluster-11 - Frontal Pole | -0.037367 (0.0342115) | -0.022933 (0.0233522)
  Brain Cluster-12 - Right Insula | -0.0549414 (0.022013) | -0.0925233 (0.0163977)
  Brain Cluster-13 - Frontal Pole | -0.1711822 (0.0322707) | -0.1896215 (0.0252413)
  Brain Cluster-14-Right Insula | -0.0592526 (0.0219242) | -0.0882445 (0.014115)

25. Secondary Outcome: Measure of Level of Anxiety
Description: The level of anxiety was assessed using the State Anxiety Inventory questionnaire. The State Anxiety Scale (S-Anxiety) evaluates the current state of anxiety. The State Anxiety Scale has 20 items. All items are rated on a 4-point scale ranging from "1 = not at all" to "4 = very much so". The scale has a minimum score of 20 and a maximum score of 80. Higher score indicates greater anxiety. State Anxiety score was measured at different time points during the study.
Time Frame: 20 minutes after arrival for study; 80, 100, & 125 minutes post drug administration
Population: Analyses included subjects who completed the behavioral study arms.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Behavioral: Drug Challenge With Methylphenidate | Behavioral: Drug Challenge With Placebo | Behavioral: Drug Challenge With Propranolol
Number analyzed (Participants) | 20 | 20 | 20
Units on a scale
  20 minutes after arrival for study | 26.35 (1.322428) | 25.7 (1.267198) | 27.65 (1.231762)
  80 minutes post drug administration | 25.75 (1.303588) | 25.5 (1.272172) | 28.3 (1.181213)
  100 minutes post drug administration | 36.4 (2.584773) | 36.2 (2.816867) | 37.9 (2.407117)
  125 minutes post drug administration | 34.15 (2.903967) | 33.25 (2.379601) | 34.31579 (2.083144)

26. Secondary Outcome: Measure of Level of Anxiety
Description: as for outcome 25
Time Frame: 20 minutes after arrival for study; 10 minutes & 145 minutes post drug administration
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 34 | 33
Units on a scale
  20 minutes after arrival for study: number analyzed (Participants) | 33 | 33
  20 minutes after arrival for study | 24.6363636 (0.9260725) | 23.1818182 (0.6099779)
  10 minutes post drug administration | 27.2352941 (1.2827241) | 24.2352941 (0.8528643)
  145 minutes post drug administration | 32.4705882 (1.3908507) | 29.6969697 (1.8512306)

27. Secondary Outcome: Measure of Heart Rate
Description: The heart rate was monitored with two disposable electrodes on the ribcage midway between the waist and the armpit.
Time Frame: 20 minutes after arrival for study; 80 minutes & 125 minutes post drug administration
Population: Analyses included subjects who completed the behavioral study arms.
Measure: Mean (Standard Error); unit: beats/minute
Arm/Group | Behavioral: Drug Challenge With Methylphenidate | Behavioral: Drug Challenge With Placebo | Behavioral: Drug Challenge With Propranolol
Number analyzed (Participants) | 20 | 20 | 20
beats/minute
  20 minutes after arrival for study | 72.8 (2.342513) | 74.35 (4.290918) | 66.35 (3.887412)
  80 minutes post drug administration | 73.6 (2.293469) | 75.1 (2.881794) | 64.6 (1.877008)
  125 minutes post drug administration | 75.75 (3.034777) | 72.45 (2.638256) | 60.05 (1.726687)

28. Secondary Outcome: Measure of Heart Rate
Description: The heart rate was monitored with two disposable electrodes on the ribcage midway between the waist and the armpit.
Time Frame: 20 minutes after arrival for study; 10 minutes & 145 minutes post drug administration
Population: Analyses included subjects who completed the fMRI study arms and had data for analysis
Measure: Mean (Standard Error); unit: beats/minute
Arm/Group | fMRI: Drug Challenge With Methylphenidate | fMRI: Drug Challenge With Placebo
Number analyzed (Participants) | 34 | 34
beats/minute
  20 minutes after arrival for study | 79.0294118 (1.4233132) | 77.2941176 (1.7900146)
  10 minutes post drug administration: number analyzed (Participants) | 33 | 34
  10 minutes post drug administration | 72.1818182 (1.4171932) | 72.6470588 (2.2260339)
  145 minutes post drug administration: number analyzed (Participants) | 33 | 34
  145 minutes post drug administration | 74.3030303 (2.3046745) | 69.7647059 (2.5201713)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Step 1/Behavioral: Drug Challenge With Methylphenidate: Participant received methylphenidate 20 mg orally during study visit
- Step 1/Behavioral: Drug Challenge With Placebo: Participant received placebo orally during study visit
- Step 1/Behavioral: Drug Challenge With Propranolol: Participants received propranolol 40mg orally during study visit
- Step 2/fMRI: Drug Challenge With Methylphenidate: Participant received methylphenidate 20 mg orally during a single day six hour study visit
- Step 2/fMRI: Drug Challenge With Placebo: Participant received placebo orally during a single day six hour study visit
Arm/Group | Step 1/Behavioral: Drug Challenge With Methylphenidate | Step 1/Behavioral: Drug Challenge With Placebo | Step 1/Behavioral: Drug Challenge With Propranolol | Step 2/fMRI: Drug Challenge With Methylphenidate | Step 2/fMRI: Drug Challenge With Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 11/20 | 10/20 | 12/20 | 0/34 | 0/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1/Behavioral: Drug Challenge With Methylphenidate (N=20) | Step 1/Behavioral: Drug Challenge With Placebo (N=20) | Step 1/Behavioral: Drug Challenge With Propranolol (N=20) | Step 2/fMRI: Drug Challenge With Methylphenidate (N=34) | Step 2/fMRI: Drug Challenge With Placebo (N=34)
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 4 | 0 | 0
Hyperhidrosis (General disorders) | 3 | 2 | 2 | 0 | 0
Irritability (General disorders) | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 8 | 6 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 2 | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 2 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT02153944/Prot_SAP_000.pdf